CLINICAL TRIAL: NCT04391283
Title: A Prospective, National, Multi-centric, Non-interventional Study of First Line Osimertinib in Chinese Patients With Locally Advanced/Metastatic，EGFR Mutation-positive NSCLC in Real World Setting
Brief Title: First Line Osimertinib for EGFR Mutation-positive Non-Small Cell Lung Cancer in Real World Chinese Setting
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: Osimertinib-RWE-01
Record Dates: First submitted 2020-04-21; First posted 2020-05-18 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Carcinoma, Non-Small-Cell Lung; Epidermal Growth Factor Receptor mutation; Osimertinib; Real World evidence; non-interventional
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood Sample Collection and Retention: about 10 mL Whole human blood samples will be collected using streck tube, sent to the NGS lab and plasma will be extracted for storage at -80℃. until test.
  Tissue Sample Collection and Retention At baseline, fresh tissue samples (or cytological samples) will be collected or 6 slices of tissue sample olefin resections obtained from surgery or 10 slices of tissue samples olefin resection obtained from puncture biopsy will be provide to central laboratory for biomarker analysis. Before tissue sample olefin resection sent to central laboratory, a pathological quality should be conducted to ensure the percentage of tumor cells is greater than 10%. Tissue sample olefin resection will be labeled and put in a box and store at room temperature
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Osimertinib — The recommended dose is 80 mg osimertinib once a day until disease progression or unacceptable toxicity according to the prescription information and clinical practice. It can be taken with or without food at the same time each day.
  Other Names: TAGRISSO

SUMMARY:
The results of phase III FLAURA study showed a significant PFS benefit for first-line Osimertinib versus standard EGFR-TKIs in patients with EGFR mutation-positive NSCLC, the median PFS was 18.9 months and 10.2 months, respectively. However, only 136 Chinese patients were enrolled in FLAURA study. The objectives of this study are to assess the efficacy and safety of Osimertinib in a real world setting in Chinese patients with locally advanced or metastatic, treatment naïve, epidermal growth factor receptor (EGFR) mutation-positive Non-Small Cell Lung Cancer (NSCLC).

DETAILED DESCRIPTION:
Total of ~30 study sites are selected for conducting this observational study. Eligible patients will be prospectively and consecutively included. Therefore, the clinical practice in the selected patients group can represent the "real-world" situation in China, and the patient's medical record will be well documented and archived in those hospitals. All data defined in the protocol will be collected during the study and entered in the Electric Data Capture (EDC), being consistent to the patients' medical records.

The most important bias of the study is that patients' characteristics will affect the treatment duration, efficacy and safety, such as, higher proportion of patients with WHO PS 2~3 enroll in the study will result in shorter TTD, poorer effectiveness and higher toxicities than expected. The ~30 sites are not randomly selected and potential selection bias exists. To minimize enrolment bias, the patients who are eligible and consent to participate in the current study will be enrolled consecutively as per protocol and without personal preference from investigators.

The self-selection bias may exit for the willingness and non-willingness participants. We'll try our best to discuss with the non-willingness participants to make sure the consistency/comparative between the willingness and non-willingness participants.

There could be a certain percentage of patients who would lost to follow up, it is unavoidable in clinical study, and is more common in real world study. We can minimize the bias by selecting the hospitals with normative and high-quality clinical practice, trying to collect the reason of lost to follow up and enhancing patient management during the follow up. The above bias is acceptable as this is a "real-world" study. Only descriptive analysis will be performed for the primary, secondary and exploratory objectives. No statistical comparisons between subgroups will be done.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent, complete all study assessments and have complete medical record;
* Histologically or cytologically documented locally advanced, metastatic NSCLC, which are not amenable to curative surgery or radiotherapy;
* With confirmation of the presence of the EGFR mutation.
* Patients must be treatment- naïve for locally advanced or metastatic NSCLC.
* Age ≥ 18 years
* Patients who plan to receive Osimertinib monotherapy as the initial first line treatment based on physician's medical judgement.

Exclusion Criteria:

* Patients who will be or were involved in any other interventional anti-tumour clinical studies for locally advanced/metastatic NSCLC currently or previously
* Any concomitant condition evaluated by physicians which is not suitable for Osimertinib treatment.
* Patients who have received the first dose of Osimertinib before the signature of ICF won't be allowed to enroll in.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with locally advanced/metastatic, EGFR mutation-positive NSCLC who are intent to be prescribed Osimertinib as the first line treatment are eligible to be the study target population.
  Base on the current clinical practice, it is estimated that the brain scans could be performed to approximately 350 patients at the baseline, approximately 200 patients' tissue or blood sample could be available at the baseline for de novo T790M analysis, and few patients with uncommon EGFR mutation, and/or patients with PS 2-3 could be included base on the current CSCO lung cancer guideline and clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Time to discontinuation (TTD) | from the date of first dose of Osimertinib in this study until the date of Osimertinib discontinuation for any reason including disease progression, treatment toxicity, death or other reason as recorded in CRF, assessed up to 36 months.
  Time to discontinuation (TTD), is defined as the time from the date of first dose of Osimertinib in this study until the date of Osimertinib discontinuation for any reason including disease progression, treatment toxicity, death or other reason as recorded in CRF. Subjects who are still on treatment at the time of analysis will be censored at the date of last dose received. Lost to follow-up patients will be censored at last documented contact with patient status "on treatment".

SECONDARY OUTCOMES:
Progression-free survival (PFS) and Progression-free survival rate (PFS rate) | from the date of first dose of Osimertinib in this study until the date of disease progression, assessed up to 36 months.
  Progression-free survival (PFS), is defined as the time from the date of first dose of Osimertinib in this study until the date of disease progression as recorded in CRF or death (by any cause in the absence of progression) regardless of whether the subject withdraws from therapy or receives another anti-cancer therapy prior to progression, which usually refer to Response Evaluation Criteria In Solid Tumours (RECIST) in clinical practice. Subjects who have not progressed or died at the time of analysis will be censored at the time of the latest date of assessment. If the subject has no evaluable visits after the baseline visit, they will be censored at 0 days unless they die before the planned visit after the baseline visit. Lost to follow-up patients who have not progressed will be censored at last documented contact with patient status "non-progression".
  Progression-free survival rate (PFS rate), is defined as the percentage of patients who do not progress on Osimertinib treatment
Objective Response Rate (ORR) and Disease Control Rate (DCR) | from the date of first dose of Osimertinib, assessed up to 6 months.
  Objective Response Rate (ORR), is defined as the percentage of patients with complete response or partial response by investigator assessment as recorded in the CRF, which usually refer to Response Evaluation Criteria In Solid Tumours (RECIST) in clinical practice.
  Disease Control Rate (DCR), is defined as the percentage of patients with non-progression by investigator assessment as recorded in the CRF, which usually refer to Response Evaluation Criteria In Solid Tumours (RECIST) in clinical practice.
Overall survival rate (OS rate) | from the date of first dose of Osimertinib in this study until the death of patients,assessed up to 48 months.
  Defined as the proportion of patients who are still alive at a particular time in the study (eg, 1 year or 2 years). The patient should be contacted 1 week after the termination of the corresponding OS analysis data to determine survival status. Lost to follow-up patients who have not progressed will be censored at last documented contact with patient status "survival".
de novo T790M mutation rate | the baseline and at the time of progression, assessed up to 36 months.
  The mutation rate of de novo T790M test by high sensitive technique (analyzed by Next Generation Sequencing platform).
  de novo T790M
Adverse events/Serious adverse events | from the date of first dose of Osimertinib in this study assessed up to 36 months.
  Incidence of Adverse Events (AEs): Nature, incidence, severity and seriousness of adverse events, Incidence of Serious Adverse Events (SAEs), which usually be graded by CTCAE v4.03 based on current clinical practice.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of College of Medicine Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goss G, Tsai CM, Shepherd FA, Bazhenova L, Lee JS, Chang GC, Crino L, Satouchi M, Chu Q, Hida T, Han JY, Juan O, Dunphy F, Nishio M, Kang JH, Majem M, Mann H, Cantarini M, Ghiorghiu S, Mitsudomi T. Osimertinib for pretreated EGFR Thr790Met-positive advanced non-small-cell lung cancer (AURA2): a multicentre, open-label, single-arm, phase 2 study. Lancet Oncol. 2016 Dec;17(12):1643-1652. doi: 10.1016/S1470-2045(16)30508-3. Epub 2016 Oct 14. PMID 27751847
- [Background] Zhou C. Lung cancer molecular epidemiology in China: recent trends. Transl Lung Cancer Res. 2014 Oct;3(5):270-9. doi: 10.3978/j.issn.2218-6751.2014.09.01. PMID 25806311
- [Background] Shi Y, Au JS, Thongprasert S, Srinivasan S, Tsai CM, Khoa MT, Heeroma K, Itoh Y, Cornelio G, Yang PC. A prospective, molecular epidemiology study of EGFR mutations in Asian patients with advanced non-small-cell lung cancer of adenocarcinoma histology (PIONEER). J Thorac Oncol. 2014 Feb;9(2):154-62. doi: 10.1097/JTO.0000000000000033. PMID 24419411
- [Background] Arcila ME, Oxnard GR, Nafa K, Riely GJ, Solomon SB, Zakowski MF, Kris MG, Pao W, Miller VA, Ladanyi M. Rebiopsy of lung cancer patients with acquired resistance to EGFR inhibitors and enhanced detection of the T790M mutation using a locked nucleic acid-based assay. Clin Cancer Res. 2011 Mar 1;17(5):1169-80. doi: 10.1158/1078-0432.CCR-10-2277. Epub 2011 Jan 19. PMID 21248300
- [Background] Jenkins S, Yang JC, Janne PA, Thress KS, Yu K, Hodge R, Weston S, Dearden S, Patel S, Cantarini M, Shepherd FA. EGFR Mutation Analysis for Prospective Patient Selection in Two Phase II Registration Studies of Osimertinib. J Thorac Oncol. 2017 Aug;12(8):1247-1256. doi: 10.1016/j.jtho.2017.05.002. Epub 2017 May 17. PMID 28527899
- [Background] John T, Akamatsu H, Delmonte A, Su WC, Lee JS, Chang GC, Huang X, Jenkins S, Wu YL. EGFR mutation analysis for prospective patient selection in AURA3 phase III trial of osimertinib versus platinum-pemetrexed in patients with EGFR T790M-positive advanced non-small-cell lung cancer. Lung Cancer. 2018 Dec;126:133-138. doi: 10.1016/j.lungcan.2018.10.027. Epub 2018 Nov 1. PMID 30527177
- [Background] Reungwetwattana T, Nakagawa K, Cho BC, Cobo M, Cho EK, Bertolini A, Bohnet S, Zhou C, Lee KH, Nogami N, Okamoto I, Leighl N, Hodge R, McKeown A, Brown AP, Rukazenkov Y, Ramalingam SS, Vansteenkiste J. CNS Response to Osimertinib Versus Standard Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitors in Patients With Untreated EGFR-Mutated Advanced Non-Small-Cell Lung Cancer. J Clin Oncol. 2018 Aug 28:JCO2018783118. doi: 10.1200/JCO.2018.78.3118. Online ahead of print. PMID 30153097
- [Background] Liu Y, Sun L, Xiong ZC, Sun X, Zhang SL, Ma JT, Han CB. Meta-analysis of the impact of de novo and acquired EGFR T790M mutations on the prognosis of patients with non-small cell lung cancer receiving EGFR-TKIs. Onco Targets Ther. 2017 Apr 24;10:2267-2279. doi: 10.2147/OTT.S133082. eCollection 2017. PMID 28479857
- [Background] Su KY, Chen HY, Li KC, Kuo ML, Yang JC, Chan WK, Ho BC, Chang GC, Shih JY, Yu SL, Yang PC. Pretreatment epidermal growth factor receptor (EGFR) T790M mutation predicts shorter EGFR tyrosine kinase inhibitor response duration in patients with non-small-cell lung cancer. J Clin Oncol. 2012 Feb 1;30(4):433-40. doi: 10.1200/JCO.2011.38.3224. Epub 2012 Jan 3. PMID 22215752
- [Result] Zheng R, Zeng H, Zhang S, Chen W. Estimates of cancer incidence and mortality in China, 2013. Chin J Cancer. 2017 Aug 17;36(1):66. doi: 10.1186/s40880-017-0234-3. PMID 28818111